CLINICAL TRIAL: NCT05105113
Title: Evaluation of Survival and Success Rates of Zirzonia Dental Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0382-19 -RMB CTIL
Record Dates: First submitted 2021-09-02; First posted 2021-11-03 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Dental Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zirconia dental implant (Experimental): Patients treated with zirconia dental implant (Tav-dental) to replace missing tooth
  Interventions: Procedure: Zirconia dental implant installation surgery

INTERVENTIONS:
Procedure: Zirconia dental implant installation surgery — Dental implant installation surgery using zirconia one-piece implant (Tav-dental)

SUMMARY:
Survival and success rates of Zirconia dental implants compared with Titanium implants (Two-Piece Zirconia implants)

DETAILED DESCRIPTION:
In the last three decades the use of dental implants to support oral rehabilitation has become a common treatment in dentistry and orthopedics.

The implants are made of titanium alloy and have shown high safety and effectiveness.

However, the gray color of the implant may be reflected through the gums and impair aesthetics in the areas of the front of the mouth.

Against this background, in recent years, implant companies have developed zirconia implants, which are white in color.

Studies have shown an aesthetic advantage for zirconia implants and zirconia structures compared to titanium when placed in an aesthetic area in patients with thin gums.

Zirconia implants are resistant to high forces and like titanium implants they undergo osteointegration into the bone, another study in dogs demonstrated an improvement in the soft and hard tissue integration in zirconia implants compared to titanium. In addition to the aesthetic benefit, zirconia implants may have an advantage in a less inflammatory response in the tissues surrounding the implant. In recent years, a number of studies have been published showing detachment of titanium particles from titanium implants which cause an inflammatory response and the absorption of supporting bone around the implant. In addition, several laboratory studies have shown an advantage for zirconia implants in terms of bacterial adsorption to the surface of the implant compared to titanium implants. Studies have been found that show higher pathogenic bacterial adsorption to titanium compared to zirconia.

TavMedical was established in 1975 and mainly specializes in the production, development and marketing of consumable medical products.

In 2011 the company began to develop dental products including implants, parts and utensils.

The company specializes mainly in zirconia dental products. Titanium implants are common and well-known implants and the company focuses its activities on promoting zirconia implants, which constitute a significant differentiation from the titanium implants currently sold in the world.

The purpose of developing zirconia dental implants is to introduce zirconia implants as a preferred alternative to the dental implants currently sold from titanium.

Also, improving the implant treatments currently offered by providing an alternative with high aesthetic results. Patients in the modern age are characterized by a high awareness of their health condition and their demand for treatment with high aesthetic results.

The natural tooth and being a metal-free material adapted to a growing trend all over the world.

Research Hypothesis - Based on the literature, the success rate and survival of zirconia implants is similar to titanium implants and stands at about 95% chance of survival.

Thus differences in the survival and success of titanium implants compared to zirconia are not expected.

Clinical inflammation markers and low-level pro-inflammatory cytokines were found around zirconia implants compared to titanium implants.

Aim of the study - Comparison of survival, success and signs of inflammation of zirconia implants compared to titanium implants.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntarily signed the informed consent form.
* Male or female patient aged ≥18 Years old.
* Replacing a missing tooth by use of implant supported restoration in implantation sites that do not require extensive augmentation procedure.
* Good primary implant stability at implant placement (35N and more).
* Compliance with study schedules and arrival at study visits.

Exclusion Criteria:

* Pregnant or lactating women.
* Imbalance diabetes.
* Head and neck rediation therapy.
* Active Periodontal disease and caries.
* Patient in need of tooth extraction and immediat implantation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate Tav- implant survival. | 12 months
  Implant survival means that implants are still in the mouth. at the time of examination, regardless of the state of the prosthesis or patient satisfaction.

SECONDARY OUTCOMES:
Evaluate Tav-Implant probing depth (IPD) | 12 months.
  refers to the distance from the gingival margin to pocket base (dental pocket).
Evaluate Tav-implant Bleeding on probe (BOP) | 12 months.
  presence or absence of bleeding of the dental pocket after probing around the implant.
Evaluate Tav-implant Gingival index (GI) changes. | 4 weeks, 12 weeks, 12 months
  Gingival index (GI) (Löe and Sillness, 1963): scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding, the score is given by visual examining the gingiva around the implant.
Evaluate Tav-implant Plaque index (PI) changes. | 4 weeks, 12 weeks, 12 months
  Plaque index (PI) (Sillness and Löe, 1964): The plaque index assesses the amount of dental plaque visible around the teeth and implants, scoring each site on 0 to 3 scale.
Evaluate Tav-implant Pink Esthetic Score (PES) changes. | 4 weeks, 12 weeks, 12 months.
  Pink Esthetic Score (PES) (Fürhauser 2005): evaluates the esthetic outcome of soft tissue around implant-supported single crowns, the score is given by visual examining the gingiva around the implant.
  A score of 2, 1, or 0 is assigned to all seven parameters. A score of 0 indicated the worst and a score of 2 indicated the best result for each variable, therefore the highest possible score of 14 denoted perfect peri-implant soft tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Zigdon, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel